CLINICAL TRIAL: NCT01664897
Title: A Pilot Phase II Study of Erlotinib for the Treatment of Patients With Refractory/Relapsed AML
Brief Title: Erlotinib Hydrochloride in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0060; NCI-2012-02073 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2012-0060 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2012-08-10; First posted 2012-08-14 (Estimated); Results first posted 2020-01-07 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2019-12

CONDITIONS: Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Adult Acute Myeloid Leukemia With Inv(16)(p13.1q22); CBFB-MYH11; Adult Acute Myeloid Leukemia With t(16;16)(p13.1;q22); CBFB-MYH11; Adult Acute Myeloid Leukemia With t(8;21); (q22; q22.1); RUNX1-RUNX1T1; Adult Acute Myeloid Leukemia With t(9;11)(p22.3;q23.3); MLLT3-KMT2A; Adult Acute Promyelocytic Leukemia With PML-RARA; Alkylating Agent-Related Acute Myeloid Leukemia; Chronic Myelomonocytic Leukemia; Myelodysplastic Syndrome; Previously Treated Myelodysplastic Syndrome; Recurrent Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelomonocytic, Acute; Leukemia, Promyelocytic, Acute; Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (erlotinib hydrochloride) (Experimental): Patients receive erlotinib hydrochloride PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Erlotinib Hydrochloride; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Erlotinib Hydrochloride — Given PO
  Other Names: Cp-358,774; OSI-774; Tarceva
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This pilot phase II trial studies how well erlotinib hydrochloride works in treating patients with relapsed or refractory acute myeloid leukemia. Erlotinib hydrochloride may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the efficacy of erlotinib (erlotinib hydrochloride) in patients with refractory or relapsed acute myeloid leukemia (AML).

II. To determine the safety and tolerability of erlotinib in this patient population.

SECONDARY OBJECTIVES:

I. To investigate inhibitory effect of this drug on spleen tyrosine kinase (SYK) and its down-stream targets such as mitogen-activated protein kinase 8 (JNK), mitogen-activated protein kinase (MAPK) and mitogen-activated protein kinase 1 (Erk).

II. To evaluate its role in janus kinase (Jak)/signal transducer and activator of transcription (STAT) pathway and to investigate erlotinib-mediated cell death and/or differentiation.

III. To quantitate concentrations of plasma erlotinib.

OUTLINE:

Patients receive erlotinib hydrochloride orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AML who have either been refractory to prior therapy or have relapsed after prior therapy; patients with myelodysplastic syndromes (MDS) or chronic myelomonocytic leukemia (CMML) who received therapy with a hypomethylating agent and progress to AML are eligible if they have received any therapy for MDS and failed (i.e., lack or loss of response) regardless of whether they have received therapy for AML or not; the World Health Organization (WHO) classification will be used for AML
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Total bilirubin =< 2 x upper limit of normal (ULN)
* Alanine aminotransferase (ALT) =< 2.5 x ULN
* Creatinine =< 2 x ULN
* Patients must provide written informed consent
* Patients must have been off chemotherapy for 2 weeks prior to entering this study, unless there is evidence of rapidly progressive disease, and must have recovered from the clinically significant toxic effects of that therapy to at least grade 1; use of hydroxyurea for patients with rapidly proliferative disease is allowed before the start of study therapy and for the first four weeks on therapy
* Patients-both males and females-with reproductive potential (i.e., menopausal for less than 1 year and not surgically sterilized) must practice effective contraceptive measures throughout the study; women of childbearing potential must provide a negative pregnancy test (serum or urine) within 14 days prior to initiation of study

Exclusion Criteria:

* Patients with known allergy or hypersensitivity to erlotinib
* Patients with any other known disease (except carcinoma in-situ) concurrent severe and/or uncontrolled medical condition (e.g. uncontrolled diabetes; cardiovascular disease including congestive heart failure New York Heart Association [NYHA] class III or IV, myocardial infarction within 6 months, and poorly controlled hypertension; chronic renal failure; or active uncontrolled infection) which, in the opinion of the investigator could compromise participation in the study
* Patients unwilling or unable to comply with the protocol
* Significant gastrointestinal disorders that may interfere with absorption of erlotinib
* Patients who can receive a stem cell transplant within 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-05-16 (Actual); Primary Completion 2018-10-25 (Actual); Study Completion 2018-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cortes, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: May 2013 to May 2014
Period: Overall Study
Arm/Group | Treatment (Erlotinib Hydrochloride)
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Erlotinib Hydrochloride)
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 16
Age, Continuous [Median (Full Range); unit: years] | 67 [20 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 20
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Participants With a Response
Description: Overall Response is complete remission (CR) + CR with incomplete hematologic recovery (CRi) + Partial remission (PR) + Hematologic improvement (HI) + Morphologic Leukemia-Free State (MLF). (CR) is Bone marrow; </=5% blasts, no Auer rods or extramedullary disease and peripheral blood counts >/= 1.0x10^9/L Neutrophils, >/= 100x10^9/L platelets and no circulating blasts. (CRi), same as CR for bone marrow and <1.0x10^9/L neutrophils and < 100x10^9/L platelets in peripheral blood counts. PR is all CR criteria if abnormal prior to treatment except >/= 50%reduction in bone marrow blast but still > 5%. MLF is </=5% myeloblasts on bone marrow . HI response must be described by the number of positively affected cell lines..
Time Frame: Up to 3 months post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Erlotinib Hydrochloride)
Number analyzed (Participants) | 29
Participants | 3

2. Primary Outcome: Incidence of Clinically Significant, Non-hematologic Grade 3 or 4 Toxicities at Least Possibly Related to Erlotinib Hydrochloride
Description: Safety summaries will include tabulations in the form of tables and listings. The number of participants affected by treatment-emergent adverse events will be reported.
Time Frame: Up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Erlotinib Hydrochloride)
Number analyzed (Participants) | 29
Participants
  Fatigue | 10
  Diarrhea | 10
  Nausea | 8
  Rash | 7

3. Primary Outcome: Overall Survival
Description: Time from date of treatment start until date of death due to any cause or last Follow-up.
Time Frame: Up to 97 weeks
Measure: Median (Full Range); unit: Weeks
Arm/Group | Treatment (Erlotinib Hydrochloride)
Number analyzed (Participants) | 29
Weeks | 14 [2.3 to 96.9]

4. Primary Outcome: Event-free Survival
Description: Time from date of treatment start until the date of first objective documentation of disease-relapse.
Time Frame: Up to 21 weeks
Measure: Median (Full Range); unit: Weeks
Arm/Group | Treatment (Erlotinib Hydrochloride)
Number analyzed (Participants) | 29
Weeks | 5 [1.7 to 21.0]

5. Secondary Outcome: Biomarker Expressions
Description: Descriptive statistics will be used to summarize the expression of biomarkers and the concentrations of plasma erlotinib hydrochloride. The Wilcoxon rank sum test will be used to compare the expressions of biomarkers and concentrations of plasma erlotinib hydrochloride between patients with and without response.
Time Frame: Up to 30 days
Population: Samples and data required for the above outcome measure were not done, therefore we cannot report any outcomes for the above outcome measure.
Arm/Group | Treatment (Erlotinib Hydrochloride)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Treatment (Erlotinib Hydrochloride)
All-Cause Mortality (participants affected / at risk) | 6/29
Serious Adverse Events (participants affected / at risk) | 23/29
Other Adverse Events (participants affected / at risk) | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Erlotinib Hydrochloride) (N=29)
Blood and Lymphatic System disorder - other (Blood and lymphatic system disorders) | 1 (1)
Death (General disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Espohageal Ulcer (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Fever (General disorders) | 3 (3)
Hematoma (Vascular disorders) | 1 (1)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Lung Infection (Infections and infestations) | 9 (10)
Nausea (Gastrointestinal disorders) | 1 (1)
Neutropenic Fever (Infections and infestations) | 5 (8)
Oral Mucositis (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (2)
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Sepsis (Infections and infestations) | 3 (4)
Skin Infection (Skin and subcutaneous tissue disorders) | 1 (1)
Thromboembolic Event (Vascular disorders) | 1 (1)
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Erlotinib Hydrochloride) (N=29)
Pneumonia (Infections and infestations) | 14 (14)
Neutropenic Fever (Infections and infestations) | 13 (13)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 11 (11)
Fatigue (General disorders) | 10 (10)
Diarrhea (Gastrointestinal disorders) | 10 (10)
Nausea (Gastrointestinal disorders) | 8 (8)
Rash (Skin and subcutaneous tissue disorders) | 7 (7)
Edema (General disorders) | 5 (5)
Muscle Aches (Musculoskeletal and connective tissue disorders) | 5 (5)
Watery eyes (Eye disorders) | 5 (5)
Dizziness (Nervous system disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-09-19): https://cdn.clinicaltrials.gov/large-docs/97/NCT01664897/Prot_SAP_000.pdf